## Feasibility of Home-based Virtual Reality Rehabilitation for the Upper Extremity in Subacute and Chronic Stroke

Statistical analysis plan

NCT03559829

March 14, 2019

Descriptive statistics (mean and standard deviation) were used to describe the primary feasibility outcome, number of days the device was used during the 8-week intervention period. Similarly, descriptive statistics were used to describe the secondary feasibility outcomes: the average daily number of minutes of device use and the user experience with the device. Changes in scores between baseline and the end of the intervention period (week 8) on the efficacy outcome measures were analyzed using paired t-tests. These efficacy outcome measures included the Jebsen-Taylor Hand Function test, the Upper Extremity Fugl-Meyer Test, the Stroke Impact Scale, and the sum of the Medical Research Council (MRC) Muscle scale score for five muscle groups (elbow flexion and extension, wrist extension, and finger flexion and extension).